CLINICAL TRIAL: NCT02306083
Title: Effect of Glucosamine on Intraocular Pressure
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Rabbani Khah, clinical professor ,ophthalmic research center, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 92182
Record Dates: First submitted 2014-09-25; First posted 2014-12-03 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2014-03

CONDITIONS: Intraocular Pressure Changes After Glucosamine Sulfate Consumption.
MeSH Terms: interventions — Economics; Glucosamine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Administration of the Placebo (Placebo Comparator): Placebo three times a day.
  Interventions: Drug: Placebo three times a day
- Administration of the glucosamine sulfate (Placebo Comparator): glucosamine sulfate 1500 mg three times a day
  Interventions: Drug: glucosamine sulfate 1500 mg three times a day

INTERVENTIONS:
Drug: Placebo three times a day
  Other Names: oral consumption
  Arms: Administration of the Placebo
Drug: glucosamine sulfate 1500 mg three times a day
  Other Names: oral consumption
  Arms: Administration of the glucosamine sulfate

SUMMARY:
In this double blind clinical trial 92 patients suffering from rheumatoid arthritis are included. Those with the history of intraocular and corneal surgery, diabetic and heavy smokers are excluded from the study. Before starting the treatment all patients undergo complete ophthalmic exam, corneal biomechanical properties assessment by Ocular Response Analyzer (ORA) and corneal thickness measurement. Patients are randomly assigned to treatment and placebo groups. Those in the treatment groups receive glucosamine sulfate 1500 mg three times a day. Those in placebo arm receive alike capsule with the same schedule. At month 3 and 6 IOP(intraocular pressure), ORA and pachymetry would be checked again.

ELIGIBILITY:
Inclusion Criteria:

* History of rheumatoid arthritis based on ACR (American College of Rheumatology)FC(functional classes).
* No history of using drugs tested in the study.

Exclusion Criteria:

* History of any kind of corneal surgery.
* History of intraocular surgery.
* History of diabetes mellitus.
* Heavy smokers.
* Unwillingness to participate in the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure changes | until 6 months
  : Goldmann applanation tonometry

SECONDARY OUTCOMES:
corneal biomechanical changes | until 6 months
  Ocular Response Analyzer (ORA)

CONTACTS AND LOCATIONS:
Locations (1):
- Islamic Republic OF Iran, Tehran, Iran